CLINICAL TRIAL: NCT02767739
Title: A Randomized Community Trial of Physical Activity Intervention in Primary Healthcare to Improve Cardiovascular Risk Factors and Health-Related Quality of Life in Older Adults
Brief Title: Effects of Physical Activity on Cardiovascular Risk and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Victoria Arija Val, Phd, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P11/67
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases; Quality of Life
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical, social and cultural activities (Experimental): Physical Activity: The training program will be supervised by a physical activity specialist and will consiste of two aerobic exercise sessions per week, including walking and stretching exercises after walking. Each session will be 60 minutes and the size of groups will be from 15 to 30 participants. Additionally, participants will receive advice about the health benefits of PA and PHC nurses using different strategies to encourage the adherence of participants to the program.
  Social and cultural support activities. Activities will include: visits to museums and libraries, cultural exhibitions, tourist attractions and dance lessons. These activities will be performed once a month.
  Interventions: Behavioral: Physical, social and cultural activities
- Control Group (No Intervention): No intervention. We will measure the variables at the begining and after 9 months.

INTERVENTIONS:
Behavioral: Physical, social and cultural activities — This intervention included two 60-min aerobic exercise sessions per week. Each session was supervised by a physical activity specialist and walking and stretching exercises were performed after programmed exercise sessions. PHC nurses were prepared to advise patients about the health benefits of PA and used different strategies to encourage the adherence of participants to the program. In addition, social and cultural support activities were included in this intervention program. These activities were performed once a month and they included: visits to museums and libraries, cultural exhibitions, tourist attractions and dance lessons.
  Arms: Physical, social and cultural activities

SUMMARY:
Community intervention trial, randomized, to promote regular PA and social and cultural support activities for 9 months in older-adult primary care users and assess their effects on cardiovascular risk factors and health-related quality of life.

DETAILED DESCRIPTION:
A structured program to promote Physical , according to the recommended guidelines and supervised by healthcare personnel should be deployed to assess their short, medium and long-term effects on CVD risk and Qulity of life. The aim of this study was to evaluate the effectiveness of a program to promote Physical, social and cultural activities for 9 months on cardiovascular risk factors and quality of life among older-adults,

ELIGIBILITY:
Inclusion Criteria:

* Adults users of 4 Primary Health Care Centers in Catalunya.

Exclusion Criteria:

* Previous episode of ischemic heart disease (<6 months).
* Outbreak of arthritis with limited ability to ambulate.
* Lung or heart disease with dyspnea mild-moderate efforts.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Physical activity level | At the begining of the intervention and after 9 months.
  It will assess at baseline and final by using the short form of the International Physical Activity Questionnarie (IPAQ-S) validated in the Catalan population. It provides a self-estimated number of hours dedicated to PA. The categories are: low, moderate and vigorous physical activity. IPAQ data will use to measure the total weekly Physical Activity level in metabolic equivalents (METs)/min/week by weighting time spent in each activity intensity level with an estimated metabolic equivalent (MET) energy expenditure
Cardiovascular risk. | At the begining of the intervention and after 9 months
  All participants will be asked if they have ever been diagnosed of hypertension, type 2 diabetes, dyslipidemia, overweight or obesity. Blood pressure will be measured with a sphygmomanometer after participants have been sitting quietly for at least five minutes; three recordings will be taken and the average of the second and third readings will be use. The cardiovascular risk will be calculated for each participant using the REGICOR scale based on Framingham criteria standardized for the Spanish population .
Biochemical analysis. | At the begining of the intervention and after 9 months.
  The biochemical parameters to analyze will be: Triglycerides, total cholesterol, HDL- and LDL-cholesterol; glycated hemoglobin and glucose. A unique study profile has been created to analyze all these parameters at the Tarraco laboratory (ISO9001:2000 certified ICS Tarragona laboratory). Blood will be extracted by PHC nurses from the fasting users in the corresponding PCC at 8:00 am. The same professional will take it to the central laboratory using the standard sample transport procedure between PCC and the central laboratory.
Antropometric measurements. | At the begining of the intervention and after 9 months.
  Weight (kg) will be measured using a balance scale with the measurement taken to the nearest 0.1 kg. Height (cm) will be measured using a balance scale with the measurement taken to the nearest 1 cm. Weight and Height measurements will be then used to calculate the body mass index [BMI: Weight (kg)/ (Height) 2 (m2)]. Waist circumference (WC), will be measured finding the top of their hip bone and the bottom of their ribs. Threfore, the tape measure will be placed in the middle between these points and wrapped around the waist.
Frequency of food consumption | At the begining of the intervention and after 9 months.
  We will use a validated food frequency questionnaire to assess food consumption. Participants will be asked to report the number of times per week or month that certain foods will be consumed (45-items). Foods will be grouped according to their nutrient composition: dairy (milk, yogurt, dairy desserts, cheese); meat/fish/eggs (red, white, processed meat and cold meat, lean, fatty fish and shellfish); total cereals (rice, pasta, bread, breakfast cereals, legumes -all type-, chocolate, biscuits, pastries and candies); fruits/vegetables (salad, tomatoes; vegetables side dish: aubergine, courgette, mushrooms; green beans, chards, spinaches, fresh fruits and canned fruits); oils and beverages (sweetened beverages, fermented beverages and alcoholic beverages), then the amount of g/day of each item will be calculated from the ECA-REF study's reference values.
Health related quality of life | At the begining of the intervention and after 9 months.
  It will assess at baseline and final of the intervention with the Spanish version of the 36-item Short Form Health Survey (SF-36). It consists of 36 items used to measure health status and outcomes from the patient's point of view, including the following 8 health concepts: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health. Two summary measures, the physical component summary (PCS) and the mental component summary (MCS), are derived from the last 8 health scores. Participant responses to each item gave a total numerical score which will transform to 0-100 scale, so that a higher score corresponds to a better health status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arija V, Villalobos F, Pedret R, Vinuesa A, Jovani D, Pascual G, Basora J. Physical activity, cardiovascular health, quality of life and blood pressure control in hypertensive subjects: randomized clinical trial. Health Qual Life Outcomes. 2018 Sep 14;16(1):184. doi: 10.1186/s12955-018-1008-6. PMID 30217193
- [Derived] Arija V, Villalobos F, Pedret R, Vinuesa A, Timon M, Basora T, Aguas D, Basora J; Pas-a-Pas research group. Effectiveness of a physical activity program on cardiovascular disease risk in adult primary health-care users: the "Pas-a-Pas" community intervention trial. BMC Public Health. 2017 Jun 15;17(1):576. doi: 10.1186/s12889-017-4485-3. PMID 28619115